CLINICAL TRIAL: NCT06123273
Title: The Effect of Exercise-Oriented Training on Physical Activity Level and Exercise Awareness in Overweight and Obese Women: A Randomized-Controlled Trial
Brief Title: The Effect of Exercise-Oriented Training on Physical Activity Level and Exercise Awareness in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Cayir, Head of Department of Family Medicine, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTU-2021-9585
Record Dates: First submitted 2023-09-05; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Overweight; Physical Inactivity
MeSH Terms: conditions — Obesity; Overweight; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group was given an exercise-oriented training
  Interventions: Behavioral: Exercise-oriented training
- Control group (No Intervention): The control group was given only routine recommendations

INTERVENTIONS:
Behavioral: Exercise-oriented training — IG received an exercise-oriented training with a 20-minute presentation including graphics, in line with clinical guidelines, in addition to routine recommendations. The training included information about the benefits of exercise and the harms of a sedentary life, the relationship between exercise and chronic diseases, suggestions to have a more active lifestyle and on how to exercise, the duration and form of exercise necessary for a healthy life, and the things to be considered while exercising. During the three-month follow-up, the subjects in the IG were called every two weeks to ask about their weight measurements, their level of exercise, and how much they walked. The subjects' questions, if any, were answered, and the interview was completed by making exercise suggestions.
  Other Names: close follow-up
  Arms: Intervention group

SUMMARY:
This study aimed to investigate the effect of an exercise-oriented training on physical activity level and exercise awareness in overweight and obese women. Participants will randomized into intervention group (IG) and control group (CG) and followed-up for three months. The International Physical Activity Questionnaire Short Form (IPAQ) will be applied to both groups at the beginning and end of the study to determine the level of physical activity, and the Exercise Health Belief Model Scale (EHBM) will be applied to evaluate the exercise awareness level, and anthropometric measurements (weight, body mass index, waist circumference) will recorded. The CG will receive no other interventions other than routine recommendations. The IG will be given face-to-face training to increase exercise awareness along with routine recommendations after the first meeting, and they will be contacted by phone every two weeks for three months.

DETAILED DESCRIPTION:
Obesity and insufficient physical activity are among the most important health problems of today. Both obesity and physical inactivity are risk factors for many chronic diseases. This study aimed to investigate the effect of an exercise-oriented training on physical activity level and exercise awareness in overweight and obese women. Participants (n=112) were randomized into intervention group (IG) and control group (CG) and followed-up for three months. The International Physical Activity Questionnaire Short Form (IPAQ) was applied to both groups at the beginning and end of the study to determine the level of physical activity, and the Exercise Health Belief Model Scale (EHBM) was applied to evaluate the exercise awareness level, and anthropometric measurements (weight, body mass index, waist circumference) were recorded. The CG received no other interventions other than routine recommendations. The IG was given face-to-face training to increase exercise awareness along with routine recommendations after the first meeting, and they were contacted by phone every two weeks for three months.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-34.9 g/m2
* Female
* Turkish

Exclusion Criteria:

* Individuals with disabilities to exercise
* pregnant/breastfeeding women
* Individuals with Stage 2-3 obesity (BMI >35 kg/m2)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female obese participants were enrolled
Enrollment: 112 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
The International Physical Activity Questionnaire Short Form was used to determine the physical activity level at the beginning and end of the study | 3 months
  The International Physical Activity Questionnaire Short Form was used to determine the physical activity level at the beginning and end of the study. The minimum score is <600 Maximal Exercise Test (MET) -minute/week while the maximum score is >3000 MET-minute/week . High score means high exercise belief.

SECONDARY OUTCOMES:
Exercise Health Belief Model Scale | 3 months
  Exercise Health Belief Model Scale was used to evaluate the exercise awareness levels of all participants. The minimum score is 25 while the maximum score is 125. High score means high exercise belief.
Anthropometric measure | 3 months
  Body Mass Index was used as an anthropometric measurement. All of the participants were recorded . It is measured as weight in kilograms divided by height in meters squared.
Body fat | 3 months
  body fat percentage were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zehranur Kacar, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No